CLINICAL TRIAL: NCT02563054
Title: An Open-Label Randomized International Multi-Center Phase III Study of Capecitabine (Xeloda) in Combination With Cisplatin Versus FU/Cisplatin in Patients With Advanced and/or Metastatic Gastric Cancer
Brief Title: A Study of Capecitabine (Xeloda) in Participants With Advanced or Metastatic Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML17032
Record Dates: First submitted 2015-09-28; First posted 2015-09-29 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Fluorouracil; Capecitabine; Cisplatin

ARMS (2):
- 5-Fluorouracil + Cisplatin (Active Comparator): Participants will receive 5-FU in combination with cisplatin upto disease progression.
  Interventions: Drug: 5-Fluorouracil; Drug: Cisplatin
- Capecitabine + Cisplatin (Experimental): Participants will receive capecitabine in combination with cisplatin upto disease progression.
  Interventions: Drug: Capecitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: 5-Fluorouracil — Participants will receive 5-FU, 800 milligrams per meter-squared (mg/m^2) per day via IV infusion during Days 1 to 5 of each 3-week cycle, for a total of 6 cycles in combination with cisplatin or upto disease progression.
  Arms: 5-Fluorouracil + Cisplatin
Drug: Capecitabine — Participants will receive oral capecitabine, 1000 mg/m^2 twice daily on Days 1 to 14 of each 3-week cycle, for a total of 6 cycles in combination with cisplatin or upto disease progression.
  Arms: Capecitabine + Cisplatin
Drug: Cisplatin — Participants will receive cisplastin, 80 mg/m^2 via IV infusion on Day 1 of each 3-week cycle, for a total of 6 cycles or upto disease progression in combination with either capecitabine or 5-FU.

SUMMARY:
This study will evaluate the efficacy and safety of oral capecitabine (Xeloda) versus 5-fluorouracil (5-FU), in combination with intravenous (IV) cisplatin, in participants with advanced and/or metastatic gastric cancer. The anticipated time on study treatment is at least 6 weeks and continued up to disease progression, and the target sample size is 300 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 to 75 years of age
* Advanced and/or metastatic gastric cancer with at least 1 measurable lesion

Exclusion Criteria:

* Uncontrolled infection
* Evidence of central nervous system (CNS) metastases
* History of other malignancy within the last 5 years, except cured basal cell cancer of the skin or cured in-situ cancer of the uterine cervix
* Radiation therapy or major surgery within 4 weeks of study drug
* Previous chemotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2003-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Time to disease progression | Up to approximately 7.3 years

SECONDARY OUTCOMES:
Objective tumor response rate | Up to approximately 7.3 years
Overall survival | Up to approximately 7.3 years
Duration of response | Up to approximately 7.3 years
Time to response | Up to approximately 7.3 years
Incidence of adverse events | Up to approximately 7.3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (34):
- Argentina (2):
  - Buenos Aires
  - Rosario
- Tegucigalpa, Belize
- Brazil (7):
  - Barretos
  - Curitiba
  - Florianópolis
  - Fortaleza
  - Porto Alegre
  - São Paulo
  - Sorocaba
- China (9):
  - Beijing
  - Guangdong
  - Hubei
  - Jiangsu
  - Jiangxi
  - Shandong
  - Shanghai
  - Suzhou
  - Tianjin
- Bogotá, Colombia
- Guatemala City, Guatemala
- Hong Kong, Hong Kong
- Kuala Lumpur, Malaysia
- Mexico (2):
  - Mexico City
  - Mérida
- Panama City, Panama
- Peru (2):
  - Callao
  - Lima
- Russia (4):
  - Kazan'
  - Moscow
  - Saint Petersburg
  - Ufa
- Seoul, South Korea
- Montevideo, Uruguay

REFERENCES:
- [Derived] Chen J, Xiong J, Wang J, Zheng L, Gao Y, Guan Z. Capecitabine/cisplatin versus 5-fluorouracil/cisplatin in Chinese patients with advanced and metastatic gastric cancer: Re-analysis of efficacy and safety data from the ML17032 phase III clinical trial. Asia Pac J Clin Oncol. 2018 Oct;14(5):e310-e316. doi: 10.1111/ajco.12832. Epub 2018 Jan 26. PMID 29372626